CLINICAL TRIAL: NCT06498349
Title: A Randomized Controlled Trial of Bilateral Subthalamic Stimulation in Patients With Parkinson's Disease and Impulse Control Disorders
Brief Title: Bilateral Subthalamic Stimulation in PD Patients With Impulse Control Disorders - STIMPulseControl
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); Philipps University Marburg (Other); University Hospital Schleswig-Holstein (Other); Czech Technical University in Prague (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Steffen Paschen, Dr. med., University of Kiel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KKS-313
Record Dates: First submitted 2024-06-17; First posted 2024-07-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Impulse Control Disorders
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Intervention Model Description: Better personalized therapy adaptation and care for patients with behavioral disorders is possible. This is often currently not possible in routine clinical practice. The scale for primary outcome used as the main target has been tested for use and is suitable for the study purpose of monitoring ICD. We now want to examine what patients with ICD benefit most from.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBS-group (Other): Within indication and clinical routine:
  bilateral high frequency deep brain stimulation of the subthalamic nucleus combined with best medical treatment
  Interventions: Procedure: bilateral high frequency deep brainstimulation of the subthalamic nucleus combined with best medical treatment; Drug: best medical treatment (BMT): Adjustment of the dopaminergic medication and non-dopaminergic therapy customized for each patient according to the latest published Consensus Group Recommendations
- BMT-group (Other): Within indication and clinical routine:
  best medical treatment
  Interventions: Drug: best medical treatment (BMT): Adjustment of the dopaminergic medication and non-dopaminergic therapy customized for each patient according to the latest published Consensus Group Recommendations

INTERVENTIONS:
Procedure: bilateral high frequency deep brainstimulation of the subthalamic nucleus combined with best medical treatment — according to widely accepted expert consensus paper
  Other Names: best medical treatment for management of impulse control in Parkinson´s disease
  Arms: DBS-group
Drug: best medical treatment (BMT): Adjustment of the dopaminergic medication and non-dopaminergic therapy customized for each patient according to the latest published Consensus Group Recommendations — according to (Debove et al (2024), 'Management of Impulse Control and Related Disorders in Parkinson's Disease: An Expert Consensus, Mov Disord.

SUMMARY:
The focus of the study is on patients Parkinson's disease showing as well behavioral disorders that can be described as pathological and are summarized under the term impulse control disorder (ICD). Changes in behavior and also pathological disorders are a common side effect of treatment for Parkinson's disease. The goal of this academic study is to compare the effect of surgical (deep brain stimulation, DBS) treatment combined with a coordinated and adapted best medical treatment (BMT) to be compared with the effect of optimized best medical treatment (BMT) alone. The stimulation arm (DBS+BMT) as well as the medication arm (BMT only) will be monitored according to clinical routine. Participants will have to agree to be randomly assigned to either deep brain stimulation in combination with the best medical treatment (DBS group) or the best medical treatment alone (BMT group). Participants will have to come regularly according to clinical routine to the clinic and complete various questionaires and scales for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment: ≤ 70 years
2. Diagnosis of PD according to MDS clinical diagnostic criteria
3. Onset of first PD motor symptoms ≥ 4 years
4. Moderate or severe impulse control disorder or related behavioral disorders according to Ardouin, with at least 1 score greater than or equal to 3 (or at least 2 scores greater than or equal to 2) on the Ardouin behaviour scale with the following items considered to reflect ICBDs or related behaviors: pathological gambling, hypersexuality, shopping, eating, hobbyism, punding and compulsive medication use
5. MDS-UPDRS III improvement of ≥ 30% in the standardized levodopa test or classical Parkinsonian tremor at rest
6. Adaptation of medical therapy has been attempted
7. MoCA ≥ 24 in the meds on condition
8. BDI-II score < 20 in the meds on condition, or Patients with moderately severe depression with a BDI-II between 20 and 28 points, strict consideration must be made with the involvement of a psychiatrist. Patients must be willing and able to comply this.
9. Patients able to understand the study requirements and the treatment procedures
10. Written informed consent before any study-specific tests or procedures are performed

    Exclusion Criteria:
11. Surgical contraindications to undergo DBS operation
12. Ongoing severe depression (BDI-II > 28)
13. suicidal ideation (item 9 of BDI-II > 1)
14. Dementia (MoCA < 24) in the meds on condition
15. Any prior movement disorder treatments that involved intracranial surgery/ablation or intracranial device implantation
16. Any other active implanted device that is likely to interfere with the implantation or functioning of the DBS system
17. Simultaneous participation in another clinical trial targeting or potentially interfering with ICD
18. Any history of recurrent seizures or haemorrhagic stroke
19. Fertile women not using adequate contraceptive methods
20. Any terminal illness with significantly reduced life expectancy which exclude DBS implantation according to standard clinical care
21. A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception
22. Any impairment that would limit subject's ability to participate in the study and perform study procedures
23. Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Ardouin Scale of Behaviour in Parkinson's Disease (ASBPD) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups with respect to the hyperdopaminergic sub-score

SECONDARY OUTCOMES:
Questionnaire for Impulsive-Compulsive Disorders in Parkinson Disease Rating Scale (QUIP RS) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Starkstein-Apathy-Scale (SAS) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Hospital Anxiety and Depression Scale (HADS) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Beck Depression Inventory (BDI) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
suicidal item 9 of the BDI | 12 months
  safety focus on suicidal item 9 of the BDI with reference to the question for the last 2 months
Neuropsychiatric-fluctuations scale (NFS) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Young mania rating scale (YMRS) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Quality of life (PDQ-39) measured by Parkinson Disease Questionaire-39 Summary Index | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Zarit Burden Interview ( ZIB) for the change of burden assessment in caregivers using the brief version | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) (parts I-IV med on/med off and stim on/stim off; if applicable | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Marconi Dyskinesia Rating Scale | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Levodopa-equivalent/dopamine-agonist dosage (LEDD) and other medication | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Pittsburgh Sleep Quality Index (PSQI) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Safety weight monitoring (BMI control) | 12 months
  Difference of change from baseline to follow-up between the two treatment groups
Montreal Cognitive Assessment (MoCA) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Clinical Global Impression (CGI-S, Severity) (CGI-C, Change) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Patient Global Impression (PGI-S, Severity) (PGI-C, Change) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Parkinson's disease Dysarthria Compound Score (PD-DCS) (Speech assessment) | 12 months
  Difference of change (improvement) from baseline to follow-up between the two treatment groups
Adverse events | 12 months
  Reporting and analysis of adverse events: Frequency, type and severity of therapy related relevant adverse events of medication or DBS
Parkinson's disease Dysarthria Compound Score (PD-DCS) | 12 months
  An intra-group comparison will be performed between the individual patient's safety speech outcome of Parkinson's disease Dysarthria Compound Score (PD-DCS) The PD-DCS is a speech acoustic summary measure of the main speech affected domains in PD, namely monopitch, monoloudness, imprecise consonants, inappropriate silences, harsh/breathy voice, and speech timing abnormalities. Acoustic proxy measures of these perceptual speech domains can be extracted from speech using modern acoustic speech analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ines Deboves, MD, Principal Investigator — University Hospital Bern, Inselspital, Department of Neurology; Paul Krack, Prof., Principal Investigator — University Hospital Bern, Inselspital, Department of Neurology; Annabel van der Weide, MD, Principal Investigator — Amsterdam University Medical Center (UMC); Rob MA De Bie, Prof., Principal Investigator — Amsterdam University Medical Center (UMC); Daniel Weintraub, Prof., Study Chair — University of Pennsylvania, Section of Geriatric Psychiatry Philadelphia; Jan Rusz, Prof., Study Chair — Czech Technical University Prague, Electrical Engineering; Ann-Kristin Helmers, Prof., Study Chair — University Hospital Kiel,UKSH, Campus Kiel, Department of Neurosurgery; Claudio Pollo, Prof., Study Chair — University Hospital Bern, Inselspital, Department of Neurology; Rick Schuurmann, Prof., Study Chair — Amsterdam University Medical Center (UMC); Jörn Rau, Study Director — Philipps-University Marburg, Coordinating Center for Clinical (KKS); Carmen Schade-Brittinger, Study Director — Philipps-University Marburg, Coordinating Center for Clinical Trials (KKS); Kerstin Winterstein, Study Director — Philipps-University Marburg, Coordinating Center for Clinical Trials (KKS)
Locations (12):
- Germany (9):
  - University Hospital Cologne, Cologne
  - University Hospital Carl Gustav Carus, Dresden
  - University Hospital Duesseldorf, Düsseldorf
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Hospital Schleswig-Holstein (UKSH), Campus Kiel, Kiel
  - University Hospital of Giessen and Marburg (UKGM), Campus Marburg, Marburg
  - Charité Campus Mitte, Mitte
  - University Hospital Tuebingen, Tübingen
  - University Hospital Wuerzburg, Würzburg
- Amsterdam University Medical Center, Amsterdam, Netherlands
- Switzerland (2):
  - University Hospital of Bern (Inselspital), Bern
  - University Hospital Zuerich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: No